CLINICAL TRIAL: NCT07360990
Title: First Pilot RCT of Episodic-Buffer-Oriented P-CRP for Adults Complex Loss and Trauma
Brief Title: Effectiveness of a Brief Psychological Intervention (P-CRP) for Complex Trauma and Loss
Acronym: P-CRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahide Betül Baydar (Other)
Responsible Party: Sponsor-Investigator, Zahide Betül Baydar, Clinical Psychologist, Istanbul Rumeli University
Organization: Istanbul Rumeli University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-53938333-050-50007
Record Dates: First submitted 2026-01-01; First posted 2026-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Trauma and Stress Related Disorders; Grief (Traumatic Grief and Existential Grief); Stress Disorder - Post-traumatic (Acute)
Keywords: Early pilot randomized control trial; Complex loss and trauma; Episodic buffer; P-CRP; Brief intervention
MeSH Terms: conditions — Trauma and Stressor Related Disorders; Prolonged Grief Disorder; Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The study is a three-arm pilot randomized controlled trial consisting of an intervention group, a control group, and a waiting-list group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psychological-cognitive reprocessing procedure (P-CRP). (Experimental): The P-CRP was the experimental group receiving four session the intervention. The Psychological-Cognitive Reprocessing Procedure (P-CRP) is a brief and a neuro-psychological intervention based on the episodic buffer model. This process facilitates the separation of cognitions from automatic processing and pulls traumatic fragments into the episodic buffer through simultaneous neuronal firing. This integration helps resolve the semantic fragmentation caused by trauma, allowing for cognitive reintegration and meaning making.
  Interventions: Behavioral: Psychological-cognitive reprocessing procedure (P-CRP).
- Expressive Narrative and Symbolic Drawing (ENSD) (Active Comparator): Control participants received four session a narrative-based expressive and symbolic drawing protocol. The intervention delivered to the control group can be characterized as an active, experiential, projective, and sensory-supported approach.
  Interventions: Behavioral: Expressive Narrative and Symbolic Drawing (ENSD)
- Waitlist Group (No Intervention): Participants in this group did not receive any active psychological intervention during the study period. They completed the pre-test and follow-up assessments at the same time intervals as the intervention groups. Following the completion of the follow-up phase, participants in the wait-list group were offered a psychological intervention protocol based on the study's findings to ensure ethical treatment standards.

INTERVENTIONS:
Behavioral: Psychological-cognitive reprocessing procedure (P-CRP). — Unlike traditional approaches, the traumatic imagery is not directly targeted in the first session. The intervention begins with the silent repetition of a word or phrase representing the core negative belief associated with the traumatic experience. . During each 1-minute set, bilateral stimulation (synchronized tapping on the shoulders only) is applied, allowing the client to process the traumatic material through spontaneously emerging associations selected by the mind itself. Rather than relying on external direction, the protocol activates internal self-regulation capacities. In this respect, it aims to promote semantic and symbolic reorganization, differing from classical cognitive restructuring or desensitization-based methods. The decision about which aspect of the experience will be processed or desensitized is determined by the client's own mental flow, thereby reinforcing a sense of trust in the mind's capacity despite the traumatic history.
  Arms: Psychological-cognitive reprocessing procedure (P-CRP).
Behavioral: Expressive Narrative and Symbolic Drawing (ENSD) — Following initial anamnesis and psychoeducation, clients recounted their trauma and drew a self-selected symbol of the event using their non-dominant hand. Each session involved discussing the memory and updating this symbol to facilitate indirect processing through creative expression.
  Arms: Expressive Narrative and Symbolic Drawing (ENSD)

SUMMARY:
The purpose of this retrospective study was to evaluate the effectiveness of a new psychotherapy technique called Psychological Cognitive Reprocessing Procedure (P-CRP) in treating trauma symptoms. The P-CRP intervention was developed and manualized by the principal investigator (Z.B.Baydar). Participants were randomly assigned to either the P-CRP intervention group, an active control group, or a waitlist condition. The study aimed to determine if this new method, which focused on episodic buffer processing, significantly reduced trauma-related psychological distress compared to standard approaches. Data collected during the intervention phase were analyzed to assess the efficacy of the P-CRP technique.

ELIGIBILITY:
Individuals were excluded if they had:

1. An Adverse Childhood Experiences (ACE) score greater than 7.
2. A history of psychotic disorder or bipolar disorder.
3. Current suicide risk.
4. Substance use disorder.
5. Prior therapeutic contact with the researcher.
6. A target traumatic event that had occurred more than one year earlier.
7. Not meeting clinical DSM-5 criteria for PTSD during the clinician-administered semi-structured interview, regardless of initial self-report scores.
8. Current participation in any other form of psychotherapy or psychiatric intervention.

Individuals were included if they had:

1. Meeting DSM-5 criteria for PTSD symptoms (verified by IES-R scores and clinician-led semi-structured interview).
2. Having experienced a target traumatic event or loss within the past 12 months.
3. Willingness to provide informed consent and participate in all intervention sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
The Impact of Event Scale -Revised (IES-R) | Baseline (Week 0), Post-intervention (Week 6), and Follow-up (Week 10) .
  The IES-R is a 22-item self-report scale designed to assess the psychological impact of traumatic experiences across three subdimensions: intrusion, avoidance, and hyperarousal. Items are rated on a 5-point Likert scale (0 = not at all to 4 = extremely) based on symptom frequency over the past seven days. Total scores range from 0 to 88, where higher scores indicate greater severity of post-traumatic stress symptoms. According to the literature, scores of 33 and above suggest a probable PTSD diagnosis. The Turkish adaptation was used, which demonstrated high validity and reliability.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI). | Baseline (Week 0), Post-intervention (Week 6), and Follow-up (Week 10)
  At the beginning of the scale, four demographic questions are included (name, gender, age, and occupation). The instrument uses a four-point Likert-type response format. The State Anxiety subscale consists of 20 items rated on a scale from (1) Not at all to (4) Very much so. The Trait Anxiety subscale also contains 20 items, with response options ranging from (1) Almost never to (4) Almost always. Cronbach's alpha coefficients reported in the Turkish adaptation were α = .72 for the State Anxiety subscale, α = .67 for the Trait Anxiety subscale, and α = .70 for the total scale; overall reliability values for the instrument have been reported to fall between α = .60 and α = .80.
The Body Sensations Questionnaire (BSQ). | Baseline (Week 0), Post-intervention (Week 6), and Follow-up (Week 10)
  It is a 17-item self-report measure assessing fear of bodily sensations associated with arousal and panic. Cronbach's alpha for the scale is reported as .92; in the current study, internal consistency was α = .93.
The Positive and Negative Affect Schedule (PANAS) | Baseline (Week 0), Post-intervention (Week 6), and Follow-up (Week 10)
  Scale is a 20-item scale consisting of 10 positive and 10 negative affect items. In the present study, Cronbach's alpha coefficients were α = .86 for Positive Affect and α = .82 for Negative Affect.

CONTACTS AND LOCATIONS:
Overall Officials: Zahide B. Baydar, Clinical Psychologist (Msc.), Principal Investigator — Istanbul Rumeli University
Locations (1):
- Zahide Betül Baydar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the current study are not publicly available due to participant confidentiality and ethical restrictions established in the informed consent agreement. However, de-identified data may be made available from the corresponding author ([Z.B.B]) upon reasonable request for scientific purposes.

REFERENCES:
- [Background] Whitall, J., Waller, S. M., Silver, K. H. C., & Macko, R. F. (2000). Repetitive bilateral arm training with rhythmic auditory cueing improves motor function in chronic hemiparetic stroke. Stroke, 31(10), 2390-2395. Whitall, J., Waller, S. M., Sorkin, J. D., Forrester, L. W., Macko, R. F., Hanley, D. F., & Goldberg, A. P. (2011). Bilateral and unilateral arm training improve motor function through differing neuroplastic mechanisms: A single-blinded randomized controlled trial. Neurorehabilitation and Neural Repair, 25(2), 118-129. Zainal, N., Newman, M., & Hong, R. (2019). Cross-cultural and gender invariance of transdiagnostic processes in the united states and singapore. Assessment, 28(2), 485-502.
- [Background] Van der Kolk, B. A. (2018). Beden kayıt tutar: Travmanın iyileşmesinde beyin, zihin ve beden (N. Cihanşümül Maral, Çev.). Nobel Yaşam. (Orijinal eser 2014'te yayımlandı) Webb, C. A., Derubeis, R. J., & Barber, J. P. (2010). Therapist adherence/competence and treatment outcome: A meta-analytic review. Journal of consulting and clinical psychology, 78(2), 200-211. Weiss, D. S., & Marmar, C. R. (1997). The Impact of Event Scale-Revised. In J. P. Wilson & T. M. Keane (Eds.), Assessing psychological trauma and PTSD (pp. 399-411). Guilford Press.
- [Background] Pagani, M., Di Lorenzo, G., Verardo, A. R., Nicolais, G., Monaco, L., Lauretti, G., Russo, R., Niolu, C., & Siracusano, A. (2012). Neurobiological correlates of EMDR monitoring-An EEG study. PLoS ONE, 7(9), e45753. Pagani, M., Amann, B. L., Landin-Romero, R., & Carletto, S. (2017). Eye Movement Desensitization and Reprocessing and slow wave sleep: A putative mechanism of action. Frontiers in Psychology, 8, 1935. Park, C. L. (2022). Meaning making following trauma. Frontiers in Psychology, 13:844891 Picó-Pérez, M., Fullana, M. À., Albajes-Eizagirre, A., Vega, D., Marco-Pallarés, J., Vilar, A., … & Soriano-Mas, C. (2022). Neural predictors of cognitive-behavior therapy outcome in anxiety-related disorders: a meta-analysis of task-based fmri studies. Psychological Medicine, 53(8), 3387-3395. Rank, O. (2001/2024). Doğum travması (S. Yücesoy, Çev.). Metis Yayınları. (Orijinal eser 1924'te yayımlandı.) Resick, P. A., Wachen, J. S., Mintz, J., Young-McCaughan, S., Roache, J. D., Borah, A. M., … & Peterson, A. L. (2015). A randomized clinical trial of group cognitive processing therapy compared with group present-centered therapy for ptsd among active duty military personnel.Journal of Consulting and Clinical Psychology, 83(6), 1058-1068. Shapiro, F. (2001). Eye movement desensitization and repro-cessing: Basic principles, protocols and procedures (2nd ed.).New York: Guilford Shapiro, F. (2021). Eye movement desensitization and reprocessing (EMDR) therapy: Basic principles, protocols, and procedures (3rd ed.). Guilford Press. Shiffrin, R. and Atkinson, R. (1969). Storage and retrieval processes in long-term memory.. Psychological Review, 76(2), 179-193. Schore, A. (2021). The interpersonal neurobiology of intersubjectivity. Frontiers in Psychology, 12. Silfwerbrand, L., Ogata, Y., Yoshimura, N., Koike, Y., & Gingnell, M. (2022). An fMRI-study of leading and following using rhythmic tapping. Social Neuroscience, 17(6), 558-567. Spielberger, C. D., Gorsuch, R. L.,& Lu
- [Background] Jung, C. G. (1968). The collected works of C. G. Jung: Vol. 9, Part 1. The archetypes and the collective unconscious (R. F. C. Hull, Trans.). Princeton University Press.Kazdin, A. E. (2019). Research design in clinical psychology (5th ed.). Pearson Lakoff, G. and Johnson, M. H. (2003). Metaphors we live by.. LeDoux, J. E. (1996). The emotional brain: The mysterious underpinnings of emotional life. Simon & Schuster. Lind, J. and Zumbo, B. D. (1993). The continuity principle in psychological research: an introduction to robust statistics.. Canadian Psychology / Psychologie Canadienne, 34(4), 407-414. Malmberg, K. J., Raaijmakers, J. G. W., & Shiffrin, R. M. (2019). 50 years of research sparked by atkinson and shiffrin (1968). Memory & Cognition, 47(4), 561-574. McEvoy, P., Nathan, P., & Norton, P. (2009). Efficacy of transdiagnostic treatments: a review of published outcome studies and future research directions. Journal of Cognitive Psychotherapy, 23(1), 20-33. Nechvatal, J. M. and Lyons, D. M. (2013). Coping changes the brain. Frontiers in Behavioral Neuroscience, 7.
- [Background] Husabø, E., Haugland, B. S. M., McLeod, B. D., Baste, V., Haaland, V. Ø., Bjaastad, J. F., … & Wergeland, G. J. (2021). Treatment fidelity in brief versus standard-length school-based interventions for youth with anxiety. School Mental Health, 14(1), 49-62.
- [Background] Foa, E. B., Huppert, J. D., & Cahill, S. P. (2006). Emotional processing theory: An update. In B. O. Rothbaum (Ed.), Pathological anxiety: Emotional processing in etiology and treatment (pp. 3 -24). Guilford Press. Gaden, T. S., Gold, C., Aßmus, J., Kvestad, I., Stordal, A. S., Bieleninik, Ł., … & Ghetti, C. (2023). Treatment fidelity in a pragmatic clinical trial of music therapy for premature infants and their parents: the longstep study. Trials, 24(1). Gazzaniga, M. S. (2000). Cerebral specialization and interhemispheric communication: Does the corpus callosum enable the human condition? Brain, 123(7), 1293-1326. Hertzog, M. (2008). Considerations in determining sample size for pilot studies. Research in Nursing & Health, 31(2), 180-191. Hinton, D. E., & Good, B. J. (2016). *Culture and PTSD: Trauma in global and historical perspective*. University of Pennsylvania Press.
- [Background] Foa EB, Kozak MJ. Emotional processing of fear: exposure to corrective information. Psychol Bull. 1986 Jan;99(1):20-35. No abstract available. PMID 2871574
- [Background] Ehlers A, Clark DM. A cognitive model of posttraumatic stress disorder. Behav Res Ther. 2000 Apr;38(4):319-45. doi: 10.1016/s0005-7967(99)00123-0. PMID 10761279
- [Background] Edwards, B. (1989). Drawing on the right side of the brain. New York: Jeremy P. Tarcher/Putnam.
- [Background] De Guio, F., St-Onge, E., Perlbarg, V., Urbain, C., Benali, H., & Cohen, L. (2012). An fMRI study comparing rhythmic finger tapping and complex movement sequences. Frontiers in Human Neuroscience, 6, 318.
- [Background] Cowan N, Elliott EM, Scott Saults J, Morey CC, Mattox S, Hismjatullina A, Conway AR. On the capacity of attention: its estimation and its role in working memory and cognitive aptitudes. Cogn Psychol. 2005 Aug;51(1):42-100. doi: 10.1016/j.cogpsych.2004.12.001. Epub 2005 Mar 2. PMID 16039935
- [Background] Brown, R. E. (2007). The life and work of Donald Olding Hebb, Canada's greatest psychologist. Proceedings of the Nova Scotian Institute of Science, 44(1), 1-25.
- [Background] Brewin CR. Episodic memory, perceptual memory, and their interaction: foundations for a theory of posttraumatic stress disorder. Psychol Bull. 2014 Jan;140(1):69-97. doi: 10.1037/a0033722. Epub 2013 Aug 5. PMID 23914721
- [Background] Bryant RA, Erlinger M, Felmingham K, Klimova A, Williams LM, Malhi G, Forbes D, Korgaonkar MS. Reappraisal-related neural predictors of treatment response to cognitive behavior therapy for post-traumatic stress disorder. Psychol Med. 2021 Oct;51(14):2454-2464. doi: 10.1017/S0033291720001129. Epub 2020 May 5. PMID 32366351
- [Background] Bonanno GA. Loss, trauma, and human resilience: have we underestimated the human capacity to thrive after extremely aversive events? Am Psychol. 2004 Jan;59(1):20-8. doi: 10.1037/0003-066X.59.1.20. PMID 14736317
- [Background] Baddeley A. The episodic buffer: a new component of working memory? Trends Cogn Sci. 2000 Nov 1;4(11):417-423. doi: 10.1016/s1364-6613(00)01538-2. PMID 11058819
- [Background] Baddeley, A. and Hitch, G. J. (1974). Working memory. Psychology of Learning and Motivation, 47-89.
- [Background] Yıldız, D. (2014). Geçerlik ve güvenirlik çalışmaları. In A. Öztürk (Ed.), Psikolojik Değerlendirme Araçları (pp. 240-260). Nobel Yayıncılık.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Ulukal, M., Demir, F., & Yalçın, M. (2013). Çocukluk Çağı Olumsuz Yaşantılar Ölçeği'nin Türkçe uyarlaması. [Bildiri/rapor].
- [Background] Spielberger, C. D., Gorsuch, R. L.,& Lushene, R. E.(1970). Manual for the State-Trait Anxiety Inventory. Consulting Psychologists Press.
- [Background] Kart, A., & Türkçapar, H. (2014). Beden Duyumları Ölçeği Türkçe formunun geçerlilik ve güvenilirlik çalışması. Klinik Psikiyatri Dergisi, 17(suppl 1), 28-37.
- [Background] Julious, S. A. (2005). Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics, 4(4), 287-291. https://doi.org/10.1002/pst.185
- [Background] Horowitz M, Wilner N, Alvarez W. Impact of Event Scale: a measure of subjective stress. Psychosom Med. 1979 May;41(3):209-18. doi: 10.1097/00006842-197905000-00004. PMID 472086
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Gündüz, A., Yaşar, A. B., Gündoğmuş, İ., Savran, C., & Konuk, E. (2018). Çocukluk Çağı Olumsuz Yaşantılar Ölçeği Türkçe Formunun geçerlilik ve güvenilirlik çalışması. Anadolu Psikiyatri Dergisi, 19(Özel sayı 1), 68-75.
- [Background] Gençöz, T. (2000).Pozitif ve Negatif Duygu Ölçeği: Geçerlik ve güvenirlik çalışması. Türk Psikoloji Dergisi, 15(46), 19-26.
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Çorapçıoğlu, A., Yargıç, İ., Geyran, P., & Kocabaşoğlu, N. (2006). Olayların Etkisi Ölçeği'nin (IES-R) Türkçe sürümünün geçerlilik ve güvenilirliği. Yeni Symposium, 44(1), 14-22.
- [Background] Creamer M, Bell R, Failla S. Psychometric properties of the Impact of Event Scale - Revised. Behav Res Ther. 2003 Dec;41(12):1489-96. doi: 10.1016/j.brat.2003.07.010. PMID 14705607
- [Background] Beck JG, Grant DM, Read JP, Clapp JD, Coffey SF, Miller LM, Palyo SA. The impact of event scale-revised: psychometric properties in a sample of motor vehicle accident survivors. J Anxiety Disord. 2008;22(2):187-98. doi: 10.1016/j.janxdis.2007.02.007. Epub 2007 Feb 24. PMID 17369016